CLINICAL TRIAL: NCT01337505
Title: An Open-Label Phase 1 Study to Investigate the Safety and Maximum Tolerated Dose of INNO-206 (Doxorubicin-6-Maleimidocaproyl Hydrazone; DOXO-EMCH) Administered as a 30 Minute Infusion Every 3 Weeks in Subjects With Advanced Solid Tumors
Brief Title: Safety and Maximum Tolerated Dose (MTD) Study of INNO-206 in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INNO-206-P1-MTD-01
Record Dates: First submitted 2011-04-14; First posted 2011-04-19 (Estimated); Last update posted 2022-02-10 (Actual); Status verified 2013-02

CONDITIONS: Malignant Solid Tumour
Keywords: INNO-206; Phase 1; DOXO-EMCH; Advanced solid tumors
MeSH Terms: interventions — DOXO-EMCH

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- INNO-206 (Experimental): INNO-206 at dosages of 230, 350, and 450 mg/m2 doxorubicin equivalents of 165, 260, and 325 mg/m2)will be administered as a 30 minute IVI on Day 1 of each cycle.
  Interventions: Drug: INNO-206

INTERVENTIONS:
Drug: INNO-206 — INNO-206 at dosages of 230, 350, and 450 mg/m2 (doxorubicin equivalents of 165, 260, and 325 mg/m2) will be administered as a 30 minute IVI on Day 1 of each cycle.
  Other Names: DOXO-EMCH

SUMMARY:
This is a phase 1b open-label study evaluating the preliminary safety and maximum tolerated dose of a new formulation of INNO-206 administered at doses of 230 mg/m2, 350 mg/m2 and 450 mg/m2 (165, 260, 325 mg/m2 doxorubicin equivalents, respectively) through intravenous infusion on Day 1 every 21 days for up to 6 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years, male or female.
* Histologically or cytologically confirmed malignant solid tumor that has relapsed or is refractory to standard therapy.
* Subjects who have received prior radiation therapy with stable CNS metastasis with no progression of brain metastasis by CT/MRI scan in last 4 weeks.
* Capable of providing informed consent and complying with trial procedures.
* ECOG performance status 0-2.
* Life expectancy >12 weeks.
* Measurable or evaluable disease according to RECIST 1.1 criteria.
* Women must not be able to become pregnant (e.g. post menopausal for at least 1 year, surgically sterile, or practicing adequate birth control methods) for the duration of the study.
* Women of child bearing potential must have a negative serum or urine pregnancy test at the Screening Visit and be non-lactating.
* Geographic accessibility to the site.

Exclusion Criteria:

* Palliative surgery, chemotherapy, immunotherapy and/or radiation less than 4 weeks prior to the Screening Visit.
* Exposure to any investigational agent within 30 days of the Screening Visit.
* Laboratory values: Screening serum creatinine greater than or equal to 1.5 mg/dL, alanine aminotransferase (ALT) greater than 3 times the upper limit of normal, total bilirubin greater than 3 times the upper limit of normal, white blood cell (WBC) count < 3500/mm3, absolute neutrophil count < 2000/mm3, platelet concentration < 100,000/mm3, hematocrit level < 33% for females or < 35% for males, or coagulation tests (PT,PTT) >1.5 times the upper limit or normal.
* Clinically evident congestive heart failure > class II of the New York Heart Association (NYHA) guidelines.
* Serious, clinically significant cardiac arrhythmias, defined as the existence of an absolute arrhythmia or ventricular arrhythmias classified as Lown III, IV or V.
* History or signs of active coronary artery disease with or without angina pectoris.
* Serious myocardial dysfunction defined scintigraphically (MUGA, myocardial scintigram)or ultrasound determined absolute left ventricular ejection fraction (LVEF) < 45% of predicted.
* History of HIV infection.
* Active, clinically significant serious infection requiring treatment with antibiotics, antivirals or antifungals.
* Major surgery within 3 weeks prior to treatment.
* Substance abuse or any condition that might interfere with the subject's participation in the study or in the evaluation of the study results.
* Any condition that is unstable and could jeopardize the subject's participation in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-04; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Safety | Up to 6 cycles (every 21 days)
  Safety will be based on adverse events, tolerability, physical examinations, vital signs, ECG results, laboratory test results. MTD: If 2 of 5 subjects an any dose level experiences a grade 3 or 4 non-hematologic toxicity, or a platelet count <25,000/uL or a neutrophil count <500/uL lasting >7 days and/or associated with fever >38.5C, 3 more subjects will be entered at that dose level. If 2 of 3 of the additional subjects experience any of the above adverse events, the dose level immediately below will be identified as the MTD.

SECONDARY OUTCOMES:
Objective response rate | Up to 6 cycles (every 21 days)
  To evaluate the objective response reate (OR; RECIST 1.1 criteria). Changes in tumor measurements from baseline values that are confirmed by repeat assessments will be assigned a status of CR or PR. OR=CR+PR.

CONTACTS AND LOCATIONS:
Overall Officials: Sant Chawla, M.D., Principal Investigator — Sarcoma Oncology Center
Locations (1):
- Sarcoma Oncology Center, Santa Monica, California, United States